CLINICAL TRIAL: NCT04634422
Title: Plasma Exchange (PLEX) and Convalescent Plasma (CCP) in COVID-19 Patients With Multiorgan Failure - the COVID PLEX+CCP Trial
Brief Title: Plasma Exchange (PLEX) and Convalescent Plasma (CCP) in COVID-19 Patients With Multiorgan Failure
Acronym: COVID-PLEX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wladimir Szpirt (Other)
Collaborators: Aalborg University Hospital (Other); Aarhus University Hospital (Other); Odense University Hospital (Other); Zealand University Hospital (Other)
Responsible Party: Sponsor-Investigator, Wladimir Szpirt, Consultant, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-20041716
Record Dates: First submitted 2020-11-14; First posted 2020-11-18 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Respiratory Failure; Renal Failure, Acute
MeSH Terms: conditions — Respiratory Insufficiency; Acute Kidney Injury | interventions — Plasma Exchange

STUDY DESIGN:
Intervention Model Description: Multicentre, parallel-grouped, stratified, centrally randomised controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plasma Exchange and convalescent Plasma (Experimental): 2 plasma exchange procedures within 24 hours and in addition 2 bags of CCP (equalling 600 ml CCP) infused at the end of the 2nd procedure.
  Interventions: Procedure: Plasma exchange and convalescent plasma
- Control without intervention (No Intervention): Standard care without the use of PLEX or convalescent plasma.

INTERVENTIONS:
Procedure: Plasma exchange and convalescent plasma — In addition to standard care, participants will receive 2 plasma exchange procedures max. 30 hours apart using the membrane or centrifuge method. PLEX will be initiated within 30 hours of randomization. The exchange volume of 60 mg of plasma per kg body weight will be substituted with albumin 5% and Ringer/saline 50% at the beginning followed by 50% FFP towards the end of the procedure. At the end of the 2nd procedure, participants will receive additional 2 units of CCP (equalling 600 ml CCP) with an administration rate of 100 to 250 ml/hr. Anticoagulation may be provided by citrate or by heparin but it is suggested that in patients with active bleeding regional citrate anticoagulation be utilized. PLEX may be performed via a central venous catheter if patient is deemed unsuitable for peripheral venous access, the latter is recommended. Possible SAE related to PLEX+CCP will be recorded as air embolism, anaphylaxis, TRALI and reported as an outcome.
  Arms: Plasma Exchange and convalescent Plasma

SUMMARY:
This Randomized Control Trial (RCT) proposes combination of extracorporeal cytokine removal by plasma exchange (PLEX) and additional infusion of convalescent plasma (CCP) collected from COVID-19 recovered individuals at the end of the PLEX procedure. The combination of cytokine removal by PLEX and CCP infusion is in onvestigators opinion more rational compared to CCP infusion alone and as such probably more effective in reducing the duration of mechanical ventilation, length of stay in the intensive care unit, and potentially also mortality.

DETAILED DESCRIPTION:
Background Severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) has caused a pandemic of coronavirus disease (COVID-19) with many patients developing severe hypoxia and some multiple organ failure. Many patients have died, and healthcare systems in several countries have been or will be overwhelmed because of a surge of patients needing hospitalisation and intensive care. There is no available proven treatment for COVID-19; the care is supportive, including respiratory, circulatory and renal support. For other patient groups with similar critical illness (acute respiratory disease syndrome and septic shock) multiple inflammatory mediators (cytokines) are linked to and probably responsible for such conditions. Thus, extracorporeal cytokine removal by plasma exchange (PLEX) has been tried in these conditions. Convalescent plasma on the other hand, may offer specific actions against SARS-CoV-2 and COVID-19. With this trial, the investigators will test the use of combined PLEX and infusion of convalescent plasma collected from COVID-19 recovered individuals at the end of the PLEX procedure in the most severely ill patients with COVID-19.

Objectives The investigators will aim to assess the effects of combination of PLEX and convalescent plasma on the number of days alive and out of hospital in adult patients with COVID-19 and multiple organ failure.

Inclusion and exclusion criteria All adult patients who have documented COVID-19 and multiple organ failure will be screened (use of respiratory and renal support). The patients who have received convalescent plasma for COVID-19, who have known hypersensitivity to plasma, who are pregnant, who the clinical team has decided not to escalate therapy, and those in whom informed consent cannot be obtained will be excluded.

Experimental intervention In addition to standard care, 2 plasma exchange procedures within 24 hours by membrane or centrifuge method. Exchange volume of 60 ml of plasma per kg of body weight with Albumin 5% in Ringer/saline as a substitution Fluid 50% at the beginning /Fresh Frozen Plasma 50% towards the end of the session and in addition 2 bags of CCP (equalling 600 ml CCP) with an administration rate of 100 to 250 ml/hr at the end of the 2nd procedure.

Control group with no intervention Standard care without the use of PLEX or convalescent plasma. Outcomes The primary outcome is days alive and out of hospital at day 90. Secondary outcomes are serious adverse events (anaphylactic reaction to CCP, new episode of septic shock or invasive fungal infection); days alive without life support at day 90; and all-cause mortality at day 28 and day 90.

Statistics Primary outcome will be compared using non-parametric statistics adjusting for the stratification variable (site). Differences will be quantified as differences in medians along with 95% confidence intervals. The mortality outcomes will be analysed using Fisher's exact test and binomial regression models with log links adjusted for the stratification variable (site) with results quantified as risk supplemented with risk differences and ratios, both with 95% confidence intervals.

Trial size Sample size calculation is based on preliminary data on days alive and out of hospital at day 90 in COVID-19 patients with multiple organ failure receiving standard of care (mean: 18 days (SD±18.36)). A sample size of n=100 per group would enable verification of a delta of 7.31 days, corresponding to a relative risk reduction of 40% with a power of 1-β = 0.80 for a two-sided t-test with α=0.05. To compensate for drop-out and sample variation a total of 110 patients are planned for inclusion in each treatment arm; i.e. 220 in total.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed SARS-CoV-2 (COVID-19) requiring intensive care AND - Use of Advanced respiratory support as Invasive mechanical ventilation OR Non-invasive ventilation or continuous use of continuous positive airway pressure (CPAP) for hypoxia OR Oxygen supplementation with an oxygen flow of at least 10 L/min independent of delivery system AND RRT (continuous or intermittent) -OR ECMO

Exclusion Criteria:

* who have received convalescent plasma for COVID-19,

  * who have known hypersensitivity to plasma,
  * who are pregnant,
  * who the clinical team has decided not to escalate therapy (except that for cardiac arrest; patients who are not for cardio-pulmonary-resuscitation may be enrolled).
  * Who have received RRT for more than 72 hours
  * Who have received mechanical ventilation for more than 14 days
  * We will not exclude patients enrolled in other interventional trials unless the protocols of the two trials collide (e.g. use of CCP by protocol). Co-enrolment agreements will be established with the sponsor/investigator to maintain an updated list of trials approved for co-enrolment (

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Alive at Day 90th | 90 days
  The primary outcome is days alive and out of hospital from randomisation to day 90.

SECONDARY OUTCOMES:
Day 8 serious adverse events | 8 days
  Serious adverse events - new episode of septic shock, anaphylactic reaction to CCP, invasive fungal infection, TACO, TRALI.
Day 28 all cause mortality | 28 days
  All-cause mortality at day 28
Days alive without life support at day 90 | 90 days
  Days alive without life support at day 90

CONTACTS AND LOCATIONS:
Overall Officials: Anders Perner, Prof, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be released after primary publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: June 30st 2024 - June 30st 2029
Access Criteria: Study Website
URL: http://www.covid-plex.com